CLINICAL TRIAL: NCT04900961
Title: Prevention and Early Treatment of the Long-term Physical Effects of Coronarvirus-19 (COVID-19): a Randomised Clinical Trial of Resistance Exercise.
Brief Title: CISCO-21 Prevent and Treat Long COVID-19.
Acronym: CISCO-21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN20CA537
Record Dates: First submitted 2021-05-10; First posted 2021-05-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Covid19
Keywords: COVID-19; Clinical trial; Graded resistance exercise; Personalised medicine; Post-COVID-19 syndrome; Long COVID
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): A personalised, resistance-based exercise intervention for patients during the convalescence phase in-hospital through to 3-months post-discharge, a duration reflecting chronic, maintenance treatment studies. To maximise enrolment of eligible patients, the intervention may be initiated in-hospital or in the community post-discharge. Resistance bands may be used according to the exercise guideline.
  Interventions: Other: Resistance Exercise
- Control (No Intervention): Standard of care treatment

INTERVENTIONS:
Other: Resistance Exercise — The exercise regimens are generic and designed not to require expert physiotherapy input, therefore, the availability of NHS physiotherapists, which may be at times limited, will not be a barrier to implementation
  Arms: Intervention

SUMMARY:
Many people have long-lasting symptoms after COVID-19, such as breathlessness, fatigue and chest pain. So far, research studies of treatments for COVID-19 have focused on the life-threatening acute illness; few studies look at treatments to improve long-term health after COVID-19. COVID-19, particularly when this requires a hospital admission, can lead to weight loss and muscle wasting, contributing to worse outcomes. Muscle strengthening (resistance-based) exercise could improve outcomes in the long-term.

DETAILED DESCRIPTION:
The rationale for our study has two main parts. The first (primary) addresses a gap in therapy, notably, for a non-pharmacological intervention. To address this gap, the investigators have set out to develop a lifestyle intervention that may be helpful to patients with persisting symptoms in the recovery (or convalescence) phase after COVID-19. Specifically, the investigators will train participants to undertake a pragmatic resistance-based exercise intervention that they can learn and apply according to their circumstances in-hospital or in the community. The rationale is predicated on providing patients with a personalised therapy option and empowering them in the self-management of their recovery following illness due to COVID-19 infection.

The second area of need is the general lack of evidence-based medicines for patients who have persisting symptoms after COVID-19. To address this gap, there is a need for rapid trials to evaluate multiple therapeutic candidates to urgently provide doctors (and their patients) with clinical evidence to inform treatment decisions. To address this gap, the investigatorsaim to create a platform for rapid trials of new treatments after COVID-19. The investigators wish to seize the opportunity afforded by this trial to set-up a transferable framework for future trials in COVID-19. The rationale is to provide a low-cost trials resource to facilitate the rapid set-up and cost-efficient delivery of multiple other trials. This will be a parallel work strand during the trial. The investigators will develop a Working Group of stakeholders from across the National Health Service (NHS) and Universities in Scotland and our COVID-19 patient and public invovlement (PPI) group (which includes co-applicants and collaborators). Key considerations include repurposing novel therapy, potential for efficacy, safety, endpoint, sample size, feasibility interim analyses, power, the Medicines and Healthcare products Regulatory Agency (MHRA) and costs. As part of the plan of work in application (Aim 3), the researchers and PPI Group will scope these potential interventions within the context of a platform trial with a view to identifying candidates to follow-on after the exercise intervention trial. This will cut the costs of doing future trials and allow more patients the opportunity to contribute to medical research that will improve outcomes for people recovering from COVID-19.

Our team is multidisciplinary, multi-ethnic, gender-balanced and drawn from across NHS Scotland, and the University of Glasgow. The investigators are leading the CISCO-19 study (ClinicalTrials.gov Identifier: NCT04403607), funded by the Chief Scientist Office (CSO), in the West of Scotland, using medical imaging of the hearts, lungs, and kidneys of patients, to understand the impact of COVID-19. The investigators have consulted with members of the public, including people with COVID-19, in designing this study.

The investigators will also undertake exploratory research into the vascular biology of COVID-19 infection. This work will be undertaken in collaboration with scientists in the University of Glasgow, including the British Heart Foundation Centre for Research Excellence and the Medical Research Council (MRC) Centre for Virus Research. A blood sample at 3 months will be collected and stored in the NHS Biorepository.

In order to assess the natural history, longer-term follow-up for health outcomes will be undertaken using electronic record linkage to patient records omitting the need for participants to undergo further research visits after the end of the trial. If after initial analysis longer term, follow up via national records is felt to be worthwhile additional funding will be sought for this.

Alignment with other national / international initiatives Our proposal will link with other prioritised studies in the United Kingdom. In general, co-enrolment would be desirable to synergise the studies. Our study will bring in new resource to enhance enrolment into existing studies, specifically, by engaging more sites, and more research staff.

ELIGIBILITY:
Patients will be classified according by clinical presentation:

A) Non-hospitalised - Positive diagnosis with persisting symptoms for at least 4 weeks from symptoms onset leading to medical review (A&E, Community COVID Hub) but not admission (Treatment group), B) Hospitalised, positive diagnosis, and with post-discharge, persistent symptoms for at least 4 weeks from symptoms onset (Treatment group), C) Hospitalised, positive diagnosis, and in convalescent phase in-hospital (Prevention group).

Groups A & B = target population for treatment of persisting symptoms post-COVID i.e. Long-COVID; Group C = Target population for prevention of Long COVID.

Inclusion Criteria:

1. Virology PCR positive laboratory diagnosis and/or point of care test positive for COVID-and/or
2. Positive Lateral Flow Test (confirmation from notes or by participant) and/or
3. Positive COVID antibody test
4. Persistent symptoms for at least 4 weeks from symptoms onset (Groups A & B only)
5. Presentation type - one of group A, B or C.

Exclusion Criteria:

1. Physiotherapy as part of standard care e.g. post intensive care unit (ICU), post high dependency unit (HDU),
2. No expectation of being able to walk within 3 months
3. Unable to provide informed consent,
4. Unable to comply with the protocol.
5. Known pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 233 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Incremental Shuttle Walk Test | at 3 months
  This is a validated measure of functional capacity, with test-retest reliability and evidence of being responsive to rehabilitation interventions.

SECONDARY OUTCOMES:
Spirometry | at 3 months
  The basic spirometry measurement will be forced vital capacity (FVC).
Handgrip Strength | at 3 months
  Handgrip strength will be recorded using a handheld dynamometer. For handgrip strength, measurements are performed until 3 measurements are within 5% of each other. Typically, 3 - 6 manoeuvres in each hand are performed. Responses in the dominant hand will be recorded.
Short Physical Performance Battery | at 3 months
  The Short Physical Performance Battery (SPPB) is a series of brief, simple physical tests including of the ability to stand for 10 seconds with the feet in 3 different positions (together side-by-side (score 0 - 1), semi-tandem (score 0 - 1), and tandem (score 0 - 2)), two timed trials of a 3m or 4m walk (fastest recorded) and the time to rise from a chair 5 times. The score ranges from 0 to 12 (higher scores reflect better extremity function). The gait and chair subtests score from 0 to 4.
EuroQol-5 dimension (EQ)-5D | at 3 months
  EuroQol-5 dimension (EQ)-5D, a patient reported outcome measure.
Patient Health Questionnaire-4 (PHQ4) | at 3 months
  Patient Health Questionnaire-4 (PHQ4), a patient reported outcome measure.
Brief Illness Perception Questionnaire (IPQ) | at 3 months
  Brief Illness Perception Questionnaire (IPQ), a patient reported outcome measure.
Duke Activity Status Index (DASI) | at 3 months
  Duke Activity Status Index (DASI), a patient reported outcome measure.
International Physical Activity Questionnaires Short Form (IPAQ-SF) | at 3 months
  International Physical Activity Questionnaires Short Form (IPAQ-SF), a patient reported outcome measure.
Fatigue questionnaire | at 3 months
  Fatigue questionnaire, a patient reported outcome measure.
Fried Frailty phenotype | 3 months
  Weight loss; exhaustion; grip strength; low physical activity; and slow walking pace
Episodes of care | at 3 months
  Episodes of healthcare care (primary, secondary, physiotherapy, rehabilitation)
Hospitalisation | at 3 months
  Hospitalisation for any reason, representing a serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, BSc MBChB PhD, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - Queen Elizabeth University Hospital, Glasgow
  - Royal Infirmary, Glasgow

IPD SHARING:
Plan to Share IPD: Undecided
The Investigator may share individual participant data (IPD) with bone fide researchers, subject to Sponsor approval.

REFERENCES:
- [Background] Guzik TJ, Mohiddin SA, Dimarco A, Patel V, Savvatis K, Marelli-Berg FM, Madhur MS, Tomaszewski M, Maffia P, D'Acquisto F, Nicklin SA, Marian AJ, Nosalski R, Murray EC, Guzik B, Berry C, Touyz RM, Kreutz R, Wang DW, Bhella D, Sagliocco O, Crea F, Thomson EC, McInnes IB. COVID-19 and the cardiovascular system: implications for risk assessment, diagnosis, and treatment options. Cardiovasc Res. 2020 Aug 1;116(10):1666-1687. doi: 10.1093/cvr/cvaa106. PMID 32352535
- [Background] Mangion K, Morrow A, Bagot C, Bayes H, Blyth KG, Church C, Corcoran D, Delles C, Gillespie L, Grieve D, Ho A, Kean S, Lang NN, Lennie V, Lowe DJ, Kellman P, Macfarlane PW, McConnachie A, Roditi G, Sykes R, Touyz RM, Sattar N, Wereski R, Wright S, Berry C. The Chief Scientist Office Cardiovascular and Pulmonary Imaging in SARS Coronavirus disease-19 (CISCO-19) study. Cardiovasc Res. 2020 Dec 1;116(14):2185-2196. doi: 10.1093/cvr/cvaa209. PMID 32702087
- [Background] Ho FK, Celis-Morales CA, Gray SR, Katikireddi SV, Niedzwiedz CL, Hastie C, Ferguson LD, Berry C, Mackay DF, Gill JM, Pell JP, Sattar N, Welsh P. Modifiable and non-modifiable risk factors for COVID-19, and comparison to risk factors for influenza and pneumonia: results from a UK Biobank prospective cohort study. BMJ Open. 2020 Nov 19;10(11):e040402. doi: 10.1136/bmjopen-2020-040402. PMID 33444201
- [Background] Briscoe M, Sykes R, Krystofiak T, Peck O, Mangion K, Berry C. Clinical significance of coronavirus disease 2019 in hospitalized patients with myocardial injury. Clin Cardiol. 2021 Mar;44(3):332-339. doi: 10.1002/clc.23530. Epub 2021 Jan 27. PMID 33501708
- [Background] Puente-Maestu L, Palange P, Casaburi R, Laveneziana P, Maltais F, Neder JA, O'Donnell DE, Onorati P, Porszasz J, Rabinovich R, Rossiter HB, Singh S, Troosters T, Ward S. Use of exercise testing in the evaluation of interventional efficacy: an official ERS statement. Eur Respir J. 2016 Feb;47(2):429-60. doi: 10.1183/13993003.00745-2015. Epub 2016 Jan 21. PMID 26797036
- [Background] Houchen-Wolloff L, Daynes E, Watt A, Chaplin E, Gardiner N, Singh S. Which functional outcome measures can we use as a surrogate for exercise capacity during remote cardiopulmonary rehabilitation assessments? A rapid narrative review. ERJ Open Res. 2020 Dec 7;6(4):00526-2020. doi: 10.1183/23120541.00526-2020. eCollection 2020 Oct. PMID 33313302
- [Background] Al Ozairi E, Alsaeed D, Taliping D, Jalali M, El Samad A, Mashankar A, Taghadom E, Guess N, Gill JMR, Sattar N, Gray C, Welsh P, Gray SR. Protocol for a randomised controlled trial to investigate the effect of home- and gym-based resistance exercise training on glycaemic control, body composition and muscle strength. Trials. 2020 Jun 22;21(1):557. doi: 10.1186/s13063-020-04480-2. PMID 32571396
- [Derived] Berry C, McKinley G, Bayes HK, Anderson D, Lang CC, Gill A, Morrow A, Sykes R, Taggart D, Kamdar A, Welsh P, Dawkes S, McConnachie A, Gray SR. Resistance Exercise Therapy After COVID-19 Infection: A Randomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2534304. doi: 10.1001/jamanetworkopen.2025.34304. PMID 41213124
- [Derived] Morrow A, Gray SR, Bayes HK, Sykes R, McGarry E, Anderson D, Boiskin D, Burke C, Cleland JGF, Goodyear C, Ibbotson T, Lang CC, McConnachie, Mair F, Mangion K, Patel M, Sattar N, Taggart D, Taylor R, Dawkes S, Berry C. Prevention and early treatment of the long-term physical effects of COVID-19 in adults: design of a randomised controlled trial of resistance exercise-CISCO-21. Trials. 2022 Aug 15;23(1):660. doi: 10.1186/s13063-022-06632-y. PMID 35971155

DOCUMENTS (1):
  • Study Protocol (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT04900961/Prot_000.pdf